CLINICAL TRIAL: NCT01792037
Title: the Effect of Single Dose of Etomidate Used During Emergency Intubation on Hemodynamics and Adrenal Cortex: a Randomized Clinical Trial
Brief Title: Single Dose of Etomidate and Adrenal Cortex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Assoc.Prof., Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 26177
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-02

CONDITIONS: Adrenocortical Deficiency; Hemodynamic Instability
MeSH Terms: interventions — Etomidate; Midazolam; Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Etomidate (Active Comparator): After taking of the blood samples, patients in Group I will be intubated with 0.3 mg/kg etomidate iv. Blood samples will be repeated in the 4th and 24th hour of the intubation.systolic, diastolic and mean arterial pressures, heart rates will be recorded with 15 minutes intervals in the first hour and after that hourly during surgery.Cortisol Levels in the 0,4th and 24th hour will be compared from the blood samples acquired.
  Interventions: Drug: Etomidate
- etomidate, steroid (Active Comparator): After taking of the blood samples, patients in Group II will be intubated with 0.3 mg/kg etomidate iv following a 2mg/kg methylprednisolone iv Blood samples will be repeated in the 4th and 24th hour of the intubation.systolic, diastolic and mean arterial pressures, heart rates will be recorded with 15 minutes intervals in the first hour and after that hourly during surgery.Cortisol Levels in the 0,4th and 24th hour will be compared from the blood samples acquired.
  Interventions: Drug: Etomidate; Drug: methylprednisolone
- midazolam (Active Comparator): After taking of the blood samples, patients in Group III will be intubated with 0.01 mg/kg midazolam iv. Blood samples will be repeated in the 4th and 24th hour of the intubation.systolic, diastolic and mean arterial pressures, heart rates will be recorded with 15 minutes intervals in the first hour and after that hourly during surgery.
  Cortisol Levels in the 0,4th and 24th hour will be compared from the blood samples acquired.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Etomidate
  Other Names: etomidate lipuro, BRAUN
  Arms: Etomidate; etomidate, steroid
Drug: Midazolam
  Other Names: Dormicum,Roche
  Arms: midazolam
Drug: methylprednisolone
  Other Names: Prednol-L, Mustafa Nevzat
  Arms: etomidate, steroid

SUMMARY:
we aim to evaluate the effects of single dose of etomidate or use of steroid prior to etomidate during emergency intubation on hemodynamics and adrenal cortex.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25-65 years old with American Society of Anesthesiology scores III or IV that have applied to emergency department and receives an indication for intubation by the intensive care unit physicians will be included to the study

Exclusion Criteria:

* Patients using steroid prior to the intubation and/or patients with chronical inflammatory diseases will be excluded from the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
effect of use of steroid on adrenal cortex prior to single dose etomidate by comparing cortisol levels | 24 hours

SECONDARY OUTCOMES:
compare effects of midazolam and etomidate on systemic blood pressure | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fatis Altindas, Prof., Study Director — Chairman of the Department of Anesthesiology
Locations (1):
- Cerrahpasa Medical Faculty Anesthesiology and Reanimation Department, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Tekwani KL, Watts HF, Sweis RT, Rzechula KH, Kulstad EB. A comparison of the effects of etomidate and midazolam on hospital length of stay in patients with suspected sepsis: a prospective, randomized study. Ann Emerg Med. 2010 Nov;56(5):481-9. doi: 10.1016/j.annemergmed.2010.05.034. Epub 2010 Sep 15. PMID 20828877